CLINICAL TRIAL: NCT00805233
Title: Combination Ranibizumab and Bromfenac for Neovascular Age-related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Peter J. Francis, MD, PhD, Oregon Health & Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF4442; eIRB4543
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2009-10

CONDITIONS: Age-Related Macular Degeneration
Keywords: Neovascular; AMD; Treatment; Lucentis; Bromfenac
MeSH Terms: conditions — Macular Degeneration | interventions — bromfenac; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Combination Ranibizumab intravitreal injection plus bromfenac ophthalmic drops
  Interventions: Drug: combination ranibizumab + bromfenac
- 2 (Active Comparator): ranibizumab injection alone.
  Interventions: Drug: ranibizumab injection alone

INTERVENTIONS:
Drug: combination ranibizumab + bromfenac — ranibizumab injection in study eye each month for 4 months then as needed each month for 8 months. Plus one drop of bromfenac in the study eye twice per day, each day, for 12 months.
  Arms: 1
Drug: ranibizumab injection alone — ranibizumab injection in study eye each month for 4 months then as needed each month for 8 months
  Arms: 2

SUMMARY:
This open-label, randomized, Phase II research study will look to see whether an investigational treatment combining bromfenac ophthalmic drops with ranibizumab intravitreal injection is safe and effective for treating wet AMD as compared to ranibizumab alone.

DETAILED DESCRIPTION:
Age Related Macular Degeneration (AMD) is the leading cause of blindness in adults over the age of 50 years. It can cause permanent loss of eyesight due to deterioration of the macula.

Ranibizumab monotherapy is currently the standard of care in neovascular AMD patients. Inflammation is believed to play an important role in AMD. Currently, MD's are investigating modulating the inflammation component of AMD with intra-ocular steroids although there is a high rate of steroid associated adverse events, such as glaucoma, cataracts and endophthalmitis.

Bromfenac is a non-steroidal anti-inflammatory drug (NSAIDS) and is currently approved for the treatment of inflammation following cataract surgery. In combination with intravitreal ranibizumab, bromfenac may also provide anti-inflammatory effects and may be a safer alternative to steroids.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 50 years
* Patients with active neovascular AMD
* If the patient has bilateral disease and qualifies for the study, both eyes may be included

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation Premenopausal women not using adequate contraception.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Current or recent participation in another simultaneous investigational drug trial may be exclusionary at the investigator's discretion
* Concurrent eye disease in the study eye that could compromise visual acuity (e.g., diabetic retinopathy, advanced glaucoma)
* Previous intravitreal steroid or anti-VEGF therapy within last 3 months.
* Patients with a concurrent corneal epithelial disruption or erosion
* Patients with immune deficiencies that would affect the ability of the cornea to heal
* Patients with a known sensitivity to any component of the formulations under investigation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Assessment of ocular adverse events, including uncontrolled inflammation, endophthalmitis, and retinal tear/detachment, abnormal sensation in eye, conjunctival hyperemia, eye irritation, eye pain, eye pruritus, eye redness, headache, and iritis | monthly

SECONDARY OUTCOMES:
Mean change in visual acuity at 3, 6 and 12 months | every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Francis, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Casey Eye Institute at Oregon Health & Science University, Portland, Oregon, United States